CLINICAL TRIAL: NCT04014465
Title: Monitoring Efficacy of Radiotherapy Based on Next Generation Sequencing Liquid Biopsy Technique in Lung Cancer and Esophageal Cancer: a Prospective Study
Brief Title: Monitoring Efficacy of Radiotherapy in Lung Cancer and Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tao Zhang, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC1923
Record Dates: First submitted 2019-07-09; First posted 2019-07-10 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Esophageal Cancer
Keywords: lung cancer; esophageal cancer; radiotherapy; ctDNA
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with radiotherapy: The patients of lung cancer or esophagueal cancer, who received definitvie RT, should included in this Cohort.

SUMMARY:
Lung cancer, one of the malignant tumors which poses a threat to human's health, has increased morbidity and mortality recently. Radiotherapy, as one of the common treatments, has important value in clinical application. Esophageal cancer, one of the most common digestive system cancers, has poor prognosis and high mortality. Esophageal cancer has high aggressive and many patients can't get surgical treatment because of the tumor metastasis at the time of diagnosis.Currently, chemoradiotherapy has become one of the standard treatment regimens for patients with unresectable esophageal cancer in National Comprehensive Cancer Network(NCCN). So radiotherapy is one of the most important treatments in esophageal cancer.

Currently, the efficacy evaluation method of radiotherapy is by imaging examination after several courses of treatment. However, new reports suggest that circulating tumor DNA(ctDNA) has the potential to be an indicator of therapeutic effectiveness and recurrence risk.

DETAILED DESCRIPTION:
Circulating free DNA (cfDNA) can be found dissolved in plasma and serum, at variable amounts. In the case of cancer patients, ctDNA is a fraction of the cfDNA derived from tumor. Currently, the ctDNA is widely used in "liquid biopsy" for not only does it carry the same somatic alterations as the tumor itself but also its percentage is correlated with tumor burden.

This study will investigate the clinical value of efficacy evaluation and prognosis of ctDNA detecting technique in patients with radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathological proved lung cancer or esophageal cancer.
* Candidate for radiotherapy.
* No history of prior anti-tumor treatment.
* Eastern Cooperative Oncology Group (ECOG) score 0,1.
* Being able to receive computed tomography (CT) and magnetic resonance imaging (MRI).
* Blood sample is available for dynamic monitoring.
* Written informed consent provided.
* Good compliance in the follow-up.

Exclusion Criteria:

* Had received radiotherapy, chemotherapy, biotherapy or other treatment that is related to lung cancer or esophageal cancer.
* The patients have the sign of any serious or uncontrolled systematic diseases that may have significant impact on the balance between risk and benefit, such as hypertension, infection of hepatitis B, hepatitis C or human immunodeficiency virus(HIV).
* With history of alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lung cancer or esophageal cancer intend to receive radiotherapy in Cancer hospital,Chinese academy of medical sciences.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 3 years
  the rate of progression free survival for 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
  the rate of overall survival for 3 years
Adverse Events | 3 years
  Number of Participants with Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen W, Zheng R, Zhang S, Zeng H, Zuo T, Xia C, Yang Z, He J. Cancer incidence and mortality in China in 2013: an analysis based on urbanization level. Chin J Cancer Res. 2017 Feb;29(1):1-10. doi: 10.21147/j.issn.1000-9604.2017.01.01. PMID 28373748
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Result] Tepper J, Krasna MJ, Niedzwiecki D, Hollis D, Reed CE, Goldberg R, Kiel K, Willett C, Sugarbaker D, Mayer R. Phase III trial of trimodality therapy with cisplatin, fluorouracil, radiotherapy, and surgery compared with surgery alone for esophageal cancer: CALGB 9781. J Clin Oncol. 2008 Mar 1;26(7):1086-92. doi: 10.1200/JCO.2007.12.9593. PMID 18309943
- [Result] Rolfo C, Castiglia M, Hong D, Alessandro R, Mertens I, Baggerman G, Zwaenepoel K, Gil-Bazo I, Passiglia F, Carreca AP, Taverna S, Vento R, Santini D, Peeters M, Russo A, Pauwels P. Liquid biopsies in lung cancer: the new ambrosia of researchers. Biochim Biophys Acta. 2014 Dec;1846(2):539-46. doi: 10.1016/j.bbcan.2014.10.001. Epub 2014 Oct 16. PMID 25444714
- [Result] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Result] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Quinn AM, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG, Swanton C. Corrigendum: Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2018 Feb 8;554(7691):264. doi: 10.1038/nature25161. Epub 2017 Dec 20. PMID 29258292
- [Derived] Wu Y, Li C, Yang Y, Zhang T, Wang J, Tang W, Li N, Bao H, Wang X, Bi N. Predicting Disease Progression in Inoperable Localized NSCLC Patients Using ctDNA Machine Learning Model. Cancer Med. 2024 Oct;13(20):e70316. doi: 10.1002/cam4.70316. PMID 39445439